CLINICAL TRIAL: NCT05007197
Title: The Effect of Diabetes Education Based on Learning Modality in Individuals With Diabetes Incompatible With Treatment on Compliance and Metabolic Goals: A Randomized Controlled Trial
Brief Title: Learning Modality in Individuals With Diabetes Incompatible
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Özlem KARDAŞ KİN, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 123456789123456789
Record Dates: First submitted 2021-08-04; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Education; Learning Style; Compliance With Treatment; Metabolic Target
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Patient Compliance

STUDY DESIGN:
Intervention Model Description: Among the individuals who applied to the outpatient clinic and were eligible for inclusion in the study, the odd numbers were assigned to the application group, and the even numbers to the control group. The practice group of 30 people and the control group were divided into 3 groups as auditory (n: 10), visual (n: 10) and physical learners (n: 10).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): After controlling the metabolic values of the individuals in the intervention group, the education were carried out according to the learning modality of the people.
  Group-specific diabetes trainings were completed in two training sessions. Each training session lasted an average of one and a half hours and a fifteen minute break was given.
  The auditory group in the intervention group, calling by phone; visual group by SMS and WhatsApp tactile group, reminder alerts were made by phone+SMS+WhatsApp.
  Interventions: Behavioral: The Effect of Diabetes Education Based on Learning Modality
- Control Group (No Intervention): The learning modality of the control group were determined and standard group training was provided with the education booklet.

INTERVENTIONS:
Behavioral: The Effect of Diabetes Education Based on Learning Modality — After controlling the metabolic values of the individuals in the intervention group, the education were carried out according to the learning modality of the people; Visual learners; education booklet, brochure, slides (enriched with pictures and videos), lecture, insulin injector-pen, glucose meters, introduction and demonstration of blood glucose tracking book Auditory learners; education booklet, slides, videos, lecture, question-answer, group work, peer group discussion, experience sharing Tactile learners; education booklet, slides, demonstration, insulin injector-pen, glucose meter doing the application of tools and equipment such as on the model, on himself, on his friend, filling in the blood glucose tracking book.
  Group-specific diabetes trainings were completed in 2 training sessions. Each training session lasted an average of 1.5 hours The learning modality of the control group were determined and standard group training was provided with the education booklet.
  Arms: Intervention Group

SUMMARY:
This study was planned to examine the effect of education based on learning styles in diabetic individuals who are incompatible with treatment, on treatment compliance and metabolic goals. The study was conducted as a randomized controlled study between January-September 2021 in Dokuz Eylül University Training and Research Hospital Endocrinology and Metabolic Diseases Polyclinic and Internal Medicine Polyclinic.

DETAILED DESCRIPTION:
Among the individuals who applied to the outpatient clinic and were eligible for inclusion in the study, the odd numbers were assigned to the application group, and the even numbers to the control group.

The practice group of 30 people and the control group were divided into 3 groups as auditory (n: 10), visual (n: 10) and physical learners (n: 10). Research data; The Individual Identification Form was collected using the Patient Compliance Scale for Type 2 DM Treatment, the BIG 16 Learning Styles Inventory, the Standardized Mini Mental Test (SMMT) and the Metabolic Goal Control Form. The training group was given according to the learning styles. The auditory group in the post-training practice group; calling by phone, to the visual group; By SMS, to the physical group; reminder alerts were made by phone + SMS. Standard training was given to the control group. Metabolic target values of the application and control groups were examined at 3 and 6 months after the training.

ELIGIBILITY:
Inclusion Criteria:

1. age range of 20-65,
2. at least 6 months diagnosis,
3. ability to communicate in Turkish,
4. mentally stable, with no vision, verbal, or hearing impairments
5. not having any obstacle to continue the implementation phase of the research (for example, pregnancy plan, change of city, etc.),
6. not having advanced hearing-vision problems and another serious disease or serious complication due to diabetes (amputation, etc.)
7. it is to get a score between 55 and 150 (incompatible with treatment) from the Patient Compliance Scale in Type 2 DM Treatment.

Exclusion Criteria:

*He/she received training on recurrent diabetes at Dokuz Eylul University Hospital.

to be,

* The patient's perception disorder and psychiatric disorder that prevent communication to be found,
* Having been diagnosed with cancer,
* Being pregnant,
* Blind retinopathy, advanced neuropathy and foot wound

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-08-28 (Estimated)

PRIMARY OUTCOMES:
Adherence to treatment | 6 months
  At the end of the education, the change in the individual's compliance with the treatment will be observed.
Physiological parameter | 6 months
  Change in metabolic targets (BMI, FBG, PBG, HDL, LDL, BP)
Effectiveness of education | 6 months
  The effect of diabetes education based on learning styles will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem KARDAS KIN, Principal Investigator — Ege UNİVERSITY
Locations (1):
- Kardaş Kin, Pazarcık, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kardas Kin O, Tureyen A. The effect of diabetes education based on learning modality in individuals with diabetes incompatible with treatment on compliance and metabolic goals: A randomized controlled trial. Prim Care Diabetes. 2022 Feb;16(1):150-155. doi: 10.1016/j.pcd.2021.12.006. Epub 2021 Dec 18. PMID 34930689